CLINICAL TRIAL: NCT02050854
Title: An Open-Label Observational Pilot Study to Evaluate the Pharmacokinetics of Aripiprazole in Subjects With Bipolar 1 Disorder or Schizophrenia Who Have a History of Suboptimal Adherence and Are Currently on Treatment With Oral Aripiprazole
Brief Title: Open-Label Observational Pilot Study to Evaluate the Pharmacokinetics of Aripiprazole in Subjects With Bipolar 1 Disorder or Schizophrenia
Status: Completed | Type: Observational
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 316-13-212
Record Dates: First submitted 2014-01-15; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Bipolar 1 Disorder; Schizophrenia; Mental Disorder; Nervous System Disorders
Keywords: Aripiprazole; Treatment Adherence
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Nervous System Diseases; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Subjects with Bipolar 1 Disorder or Schizophrenia who have a history of suboptimal adherence and are currently on treatment with oral aripiprazole

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of aripiprazole in subjects with Bipolar 1 Disorder or Schizophrenia who have a history of suboptimal aderence and are currently on treatment with oral aripiprazole.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetics of aripiprazole in subjects with Bipolar 1 Disorder or Schizophrenia who have a history of suboptimal aderence and are currently on treatment with oral aripiprazole. This will be an open-label observational pilot trial to compare the PK profile of aripiprazole at Visit 1 of subjects who are receiving oral aripiprazole and who have the potential for suboptimal adherent behavior with their assigned medication.

Information obtained in the current trial will be used to inform the conduct of a randomized, open-label, parallel-group trial to assess between-group change from baseline adherence using PK sampling in subjects receiving oral aripiprazole with or without the MIND1 System (Protocol 316-13-211).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 to 55 years of age (inclusive) at time of informed consent
* Subjects with a primary current Axis 1 disorder of bipolar 1 disorder or schizophrenia as defined by DSM-IV-TR criteria, who have been treated in the outpatient setting for at least 2 months before screening
* Subjects with a score of 1-7 on the Morisky 8-Item Medication Adherence Scale (MMAS-8)
* Subjects with bipolar 1 disorder who have a YMRS score of 10 to 25 (inclusive), or subjects with schizophrenia who have a PANSS score of 60 to 90 (inclusive)
* Subjects able to ingest oral medication
* Subjects currently prescribed oral aripiprazole for either bipolar 1 disorder or schizophrenia, and who have not had any changes in their Aripiprazole regimen or dose over the last 2 weeks
* Subjects who have an exacerbation of mood or psychotic symptoms when they are not receiving treatment or are noncompliant with treatment for their bipolar 1 disorder or schizophrenia
* For subjects enrolled with bipolar 1 disorder, the current bipolar episode is mixed or manic (the current must not be a depressive episode)

Exclusion Criteria:

* Subjects with a current Axis I (DSM-IV-TR) diagnosis other than bipolar 1 disorder or schizophrenia
* Subjects with a current Axis II (DSM-IV-TR) diagnosis
* Subjects not able to self-administer their medication
* Subjects who reside in or attend a facility where medication is administered to them
* Subjects who have a score of 0 or 8 on the Morisky 8-Item Medication Adherence Scale (MMAS-8)
* Subjects who currently meet DSM-IV-TR criteria for substance dependence
* Subjects with a history of inpatient hospitalization for any psychiatric reason within the past 2 months before screening
* Subjects who have received any investigational product within the last 30 days
* Subjects known to be allergic, intolerant, or unresponsive to prior treatment with Aripiprazole or other quinolinones
* Subjects who, per investigator's judgment, are acutely psychotic or manic and/or exhibit symptoms currently requiring hospitalization

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Mean log transformed-area under the plasma concentration-time curve (AUC) at Visit 1 for subjects receiving oral aripiprazole, compared to historical values | Visit 1 (Day 1)

SECONDARY OUTCOMES:
Potential relationships between a clinically accepted indicator of non-adherent behavior, the Morisky 8-item Medication Adherence scale (MMAS-8), and aripiprazole concentrations in subjects | Visit 1 (Day 1) to End of Study

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Largay, MD, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (5):
- United States (5):
  - Garden Grove, California
  - Atlanta, Georgia
  - Decatur, Georgia
  - Rockville, Maryland
  - Bellevue, Washington